CLINICAL TRIAL: NCT01295099
Title: Keloid Scarring:A Randomized Clinical and Laboratory Based Study on the Treatment and Differentiation Factors of the Local Disease
Brief Title: Keloid Scarring: Treatment and Pathophysiology
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KS001
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2022-10

CONDITIONS: Keloid Scar
Keywords: scar formation; 5-FU; genetic link; psychological impact; social impact
MeSH Terms: conditions — Keloid | interventions — Fluorouracil; Radiotherapy; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 5-Fluorouracil (Active Comparator): Patients with small keloidal scars to have intralesional 5FU injected
  Interventions: Drug: 5- fluorouracil
- Radiotherapy (Active Comparator): Large keloid scars undergo extralesional excision and radiotherapy
  Interventions: Radiation: radiotherapy
- TAC (Active Comparator)
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: 5- fluorouracil — 5mg of 5FU injected per 1cm square, at 6 week intervals for 30 weeks = 6 sessions
  Arms: 5-Fluorouracil
Radiation: radiotherapy — after complete excision of keloid they have a single session of radiotherapy
  Arms: Radiotherapy
Drug: Triamcinolone — TAC 10mg in 1ml injected intralesional
  Arms: TAC

SUMMARY:
To clarify the mechanisms of Keloid scar formation.

Elucidate the action and therapeutic value of 5-FU in Keloid scar treatment

Identify the genetic link with Keloid scar formation.

Quantify the psychological/social impact in keloid scarring patients

ELIGIBILITY:
Inclusion Criteria:

* Adult ( > 18 years old).
* Keloid scarring present.
* Able to understand and give informed consent.
* Patients giving informed consent to donate keloidal or non-affected skin when that is redundant after a procedure (i.e. BBR, Abdominoplasty).
* Patients with a strong familial pedigree of keloid scar formation.

Exclusion Criteria:

* Open wound at or proximity of the lesion

  * Infected lesion
  * Pregnant or planning pregnancy in the near future
  * Lactating (Breast Feeding)
  * Abnormal renal or liver function tests
  * Atrophic scars
  * Patient under 18 years of age
  * Immunocompromised
  * OR immunosuppressed

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Keloid Scar Reduction | 18 months
  Using a 3D scanner to observe the reduction of the scar volume measured in cubic centimetres

CONTACTS AND LOCATIONS:
Locations (1):
- Barts and the London NHS Trust, London, UK, United Kingdom

REFERENCES:
- See also: Related Info — http://www.keloids.co.uk